CLINICAL TRIAL: NCT02793765
Title: Docetaxel Followed by Provenge in Castration-Resistant Prostate Cancer
Brief Title: Docetaxel Followed by Provenge in Metastatic Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dendreon was sold and new company decided not to fund study.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert J Amato, Director and Professor, Department of Internal Medicine, Division of Oncology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-15-104; HSC-MS-15-0883 (Other: CPHS)
Record Dates: First submitted 2016-06-02; First posted 2016-06-08 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Advanced Prostate Cancer; Castration-Resistant Prostate Cancer; Adenocarcinoma of the prostate; Metastatic disease; CRPC
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel & Sipuleucel-T (Experimental): 75 mg/m2 docetaxel IV over 1-hour every 21 days x 6 cycles; 28 day rest then Sipuleucel-T IV over 1-hour every 14 days for 3 doses
  Interventions: Drug: Docetaxel; Biological: Sipuleucel-T

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere; Docefrez
Biological: Sipuleucel-T
  Other Names: Provenge

SUMMARY:
This clinical study will evaluate the role of combination therapy of docetaxel followed by Provenge for patients with metastatic castration-resistant prostate cancer (CRPC, (prostate cancer that is resistant to medical or surgical treatments that lower testosterone). The purpose of this study is to look at the combination therapy of docetaxel followed by Provenge to correlate the immunological biomarkers with clinical results for therapy. Biomarkers are genes, proteins and other molecules that affect how cancer cells grow, multiply, die and respond to other compounds in the body. The study drugs are approved by the Food and Drug Administration (FDA).

Treatment will be administered on an outpatient basis. Patients will receive 6 cycles of docetaxel followed by Provenge. Docetaxel is an antineoplastic (chemotherapy that affects cancer cell growth) agent. Docetaxel dose of 75 mg/m2 will be given intravenously as a 1-hour infusion every 21 days on Day 1 for 6 cycles. Provenge is an immunotherapy (vaccine made from patient's own blood cells) that reprograms immune cells to attack cancer. A course of therapy consists of three doses of Provenge administered at 2-week intervals.

The strategy aims to determine whether cytokine production and T cell infiltration of tumor cells could favor regression using a combination of chemotherapy plus vaccine. Tissue endpoints will include biopsies prior to first chemotherapy and first vaccine therapy and at the end of each therapy. Prostate cancer tissue infiltrates will be studied for expression of CD3, CD4, CD8, CD25/FOX3P, CD56, CTLA-4, PD-1, and Ki67. Additional immunological endpoints will be secondary antigen spread and various cytokine biomarkers.

DETAILED DESCRIPTION:
Castration-resistant prostate cancer (CRPC) develops serial treatment resistance and is considered incurable. It is a largely indolent disease, which would give the body time to mount an effective immune response. CRPC is therefore potentially well suited for vaccine therapy.

Docetaxel is an antineoplastic agent belonging to the taxoid family. The FDA-approved course of therapy for prostate cancer consists of 75 mg/m2 docetaxel given intravenously as a 1-hour infusion every 21 days on Day 1.

Sipuleucel-T (Provenge), is an FDA-approved cancer vaccine therapy manufactured by culturing an individual's own freshly isolated peripheral blood mononuclear cells (PBMCs), including antigen-presenting cells (APCs) and T cells, with a fusion protein (PA-2024) composed of prostatic acid phosphatase (PAP) linked to granulocyte macrophage-colony stimulating factor (GM-CSF). A course of therapy consists of three doses of Provenge administered at 2-week intervals.

This is an open-label phase II study in taxane-naïve patients with metastatic CRPC of docetaxel followed by Provenge. Adult (age >18 years) men with metastatic CRPC. pathologically-confirmed adenocarcinoma of the prostate with clinical or radiologic evidence of metastatic disease that has progressed despite treatment with anti-androgens, inhibitors of adrenal-produced androgens (abiraterone), or androgen receptor inhibitors (enzalutamide), and who, prior to study entry are candidates to receive Standard of Care chemotherapy (e.g., docetaxel/prednisone) or immunotherapy (Provenge), will be enrolled in this study.

This study will recruit a total of 32 patients with metastatic CRPC. Patients will receive 6 cycles of docetaxel followed by Provenge. Treatment will be administered on an outpatient basis. Patients must meet one of the following prognostic criteria:

* PSA doubling time ≤6 months
* >10 bone lesions (only if they meet PSA doubling time criteria)
* Visceral metastases
* Bone and lymph node lesions

The primary objective of this study is to characterize the immunological biomarkers during therapy and correlate the immunological biomarkers with clinical outcome. The strategy aims to determine whether cytokine production and T cell infiltration of tumor cells could favor regression using a combination of chemotherapy plus vaccine. Tissue endpoints will include biopsies prior to chemotherapy, on day 14 during the rest period between therapies and after vaccine therapy. Prostate cancer tissue infiltrates will be studied for expression of CD3, CD4, CD8, CD25/FOX3P, CD56, CTLA-4, PD-1, and Ki67. Additional immunological endpoints will be secondary antigen spread and various cytokine biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years and older.
* Pathologic confirmation of prostate adenocarcinoma.
* Asymptomatic or minimally symptomatic disease.
* Presence of skeletal or visceral/nodal metastasis confirmed by MRI, scintigraphy, or CT scan
* Disease progression despite androgen deprivation therapy (ADT) as indicated by:

  * PSA increase indicated by two consecutive higher values over baseline at assessments performed at least 7 days apart from each other in the previous 28 days with the absolute value ≥5 ng/ml and ≥50% above the minimum PSA reached during ADT or above the pre-treatment level, if no response was observed; OR
  * Progression of measurable lymph nodes (≥15 mm) or visceral lesion measureable per RECIST v1.1 criteria; OR
  * New bone lesions (>10 lesions total) appearing on bone scan/imaging compared with a prior scan. Bone scan to be performed at screening or within the previous 28 days.
* Maintenance of castrate conditions: Patients who have not had a surgical orchiectomy must continue with hormone therapy (GnRH/LHRH agonists or antagonists) to maintain levels of serum testosterone of <50 ng/dl.
* Patient is clinically immunocompetent. Clinical immunocompetence will be assumed unless a subject has been diagnosed as being immunosuppressed, is receiving oral steroids (nasal sprays and inhalers are permitted), is receiving immunosuppressive chemotherapy for oncologic disorders, or is receiving immunosuppressive therapy following transplant, in which case they will be excluded.
* Peripheral neuropathy grade ≤1.
* Laboratory criteria:

  * Adequate bone marrow function:

    1. White blood cells ≥4000/mm3
    2. Absolute neutrophil count ≥1500/mm3
    3. Absolute lymphocyte count ≥500/µl
    4. Hemoglobin ≥10 g/dl
    5. Platelet count ≥100,000/mm3
  * Total bilirubin within normal limits (benign hereditary hyperbilirubinemias, e.g., Gilbert's syndrome, are permitted)
  * Renal function creatinine ≤1.5 x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be within normal range.
* Life expectancy of at least 6 months based on Investigators' judgment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* At least 4 weeks after surgery or radiotherapy
* If patients have been receiving bisphosphonate or denosumab, they can continue either medication.
* Sufficient washout period from previous anti-androgen and hormonal therapies (PSA regression verification required after casodex withdrawal during the 6-week washout period).
* Patient is willing and available to attend clinic visits at least every 2 weeks.
* Signed, informed consent, including patient's ability to comprehend its contents

Exclusion Criteria:

* Patient has "currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy >5 years previously and have no known evidence of residual or recurrent disease.
* Current symptomatic cord compression requiring surgery or radiation therapy
* Prior chemotherapy for prostate cancer
* Patient is using supplements or complementary medicines/botanicals. Patients should review the label with their doctor prior to enrolment. The following exceptions are permitted at screening and during the course of the study.

  * Conventional multivitamin supplements
  * Selenium
  * Lycopene
  * Soy supplements
  * Vitamin E
  * Fish oil supplements
  * Vitamin D
  * Glucosamine supplements
  * Age-related eye disease vitamins
  * Ginkgo biloba
* Patient co-morbidities:

  * HIV positive
  * Acute hepatitis B (HBV) or active hepatitis C (HCV)
  * Clinical and laboratory evidence of active bacterial, viral, or fungal infection requiring systemic treatment
  * Clinically significant cardiovascular disease including

    1. Symptomatic congestive heart failure
    2. Unstable angina pectoris
    3. Serious cardiac arrhythmia requiring medication
    4. Uncontrolled hypertension >150/100mm Hg (if controlled with medication this is not an exclusion).
    5. Hypotension
    6. Myocardial infarct or ventricular arrhythmia or stroke within a 6-month period prior to inclusion, ejection fraction (EF) <40%, or serious cardiac conduction system disorders
    7. Patient is exhibiting evidence of symptomatic congestive heart failure, pulmonary embolus, vascular thrombosis, transient ischemic attack, cerebrovascular accident, unstable angina, myocardial infarction or active ischemia if a pacemaker is not present on electrocardiogram (ECG). An ECG must be performed at screening unless the subject has measurable disease in which case an ECG taken prior to screening but within 28 days of start of treatment will be accepted.
  * Pleural and pericardial effusion of any CTCAE grade
  * Rheumatoid disease (asymptomatic subjects with controlled and rarely flaring rheumatoid arthritis are also excluded)
  * Peripheral neuropathy having a CTCAE grade ≥2
  * History of malignant disease (with the exception of non-melanoma skin tumors) in the preceding 5 years
  * Active autoimmune disease requiring treatment (except non-insulin-dependent diabetes mellitus)
  * History of severe forms of primary immune deficiencies
  * History of anaphylaxis or other serious reactions following vaccination
  * Uncontrolled co-morbidities including psychiatric or social conditions which, in the Investigator's opinion, would prevent participation in the trial
* Patient has had major surgery or radiation therapy completed < 4 weeks prior to screening.
* Patient has had prior exposure to the radiopharmaceuticals radium 223, strontium, or samarium within 8 weeks prior to screening.
* Patient is receiving concurrent chemotherapy, immunotherapy, radiotherapy, or investigational agents.
* Patient has cerebral metastases (known from previous investigations or clinically detectable).
* Patient has serum testosterone >50 ng/dl.
* Systemic corticosteroids at doses >40 mg hydrocortisone daily or equivalent for any reason other than (a) prescribed as replacement therapy in the case of adrenal insufficiency or (b) oral dexamethasone administration used in combination with docetaxel.
* Patient has in the opinion of the physician a serious or uncontrolled intercurrent infection or non-malignant medical illness which is uncontrolled.
* Systemic immunosuppressive therapy for any reason.
* Treatment with anti-androgens, inhibitors of adrenal-produced androgens (abiraterone), androgen receptor inhibitors (enzalutamide), or other hormonal tumor-focused treatment performed on the day of screening or within the previous 4 weeks, including any dose of megestrol acetate, finasteride, any herbal product known to decrease PSA levels (e.g., saw palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to screening. Progressive disease (as defined above) must be documented after discontinuation of the therapy.
* Refusal to sign the informed consent.
* Participation in a clinical trial using experimental therapy within the last 60 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Cytokine activity | 18 months
  measured by staining assays
T-cell Proliferation | 18 months
  measured by flow cytometry
Serum Levels | 18 months
  measured by staining assays
Tissue Infiltration | 18 months
  measured by staining assays
Secondary antigen Spread | 18 months
  measured by flow cytometry

SECONDARY OUTCOMES:
Radiographic progression-free survival | 18 months
PSA Response Rate | 18 months
Time to PSA progression | 18 months
Measure CTCs and characterize response | 18 months
Objective tumor response rate | 18 months
Number of Adverse Events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No